CLINICAL TRIAL: NCT06981663
Title: Potential Effects of Fibres Combined With Probiotics on Uric Acid and Related Metabolites in an ex Vivo Fermentation Model
Brief Title: Effects of Fibres Combined With Probiotics on Uric Acid in an ex Vivo Fermentation Model
Status: Recruiting | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Julia König, PhD, Associate Professor, Örebro University, Sweden
Other Study IDs: 2025-01926-01; 2025-01926-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2025-04-30; First posted 2025-05-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hyperuricemia
Keywords: hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we will collect faecal samples from individuals with hyperuricaemia (assessed by blood test) and perform in vitro faecal fermentation studies to assess how probiotics in combination with fibres affect urate metabolism in these faecal samples.

DETAILED DESCRIPTION:
In this study, the investigators will collect blood samples to check if recruited participants have hyperuricemia, and if yes, stool samples will be collected for laboratory faecal fermentation tests. The research project aims to investigate the effects of probiotics and dietary fibers on stool samples, to understand if and how they can support the gut microbiota to break down uric acid in the gut.

Participation in the study involves data collection and sampling on three occasions. During the first visit, participants will provide a blood sample, and if they have increased urate levels, they will be asked to complete questionnaires and be provided with materials for stool sampling during the second visit. During the third visit, they will provide the stool sample, which will then be used in the faecal fermentation experiments, where different fibres (beta-glucans) will be tested in combination with probiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedures
2. Age 18-80 years old
3. BMI range 18.5-35 kg/m2
4. Blood uric acid above 0.36 mmol/L (6 mg/dl)
5. Willing to abstain from regular consumption of probiotic supplements or food products containing probiotic bacteria (including fermented food and beverages), until collection of faecal material
6. Willing to abstain from regular consumption of supplements and medications known to alter gastrointestinal function or inflammatory status during the study, until collection of faecal material

Exclusion Criteria:

1. Diagnosis of type 1 and/or type 2 diabetes
2. Diagnosed inflammatory bowel disease (IBD)
3. Current diagnosis of psychiatric disease/s or syndromes
4. Current diagnosis of neurodegenerative disease
5. Current pregnancy or breastfeeding
6. History of complicated gastrointestinal surgery
7. Systemic use of antibiotics and/or steroid medication in the last 4 months prior to inclusion
8. Regular use of any non-steroidal anti-inflammatory drug (NSAID) for the last 2 months
9. Consumption of any NSAID within 3 days of sample collection
10. Current (or within the last 4 weeks prior to study start) use of probiotic supplementation
11. Any condition or intake of medication which could substantially interfere with the outcome of the study, as decided by the principal investigator's discretion
12. After being included in the study and until collection of faecal material, starting any medication or treatment that could potentially influence the study participation and/or study analysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hyperuricaemic adults
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Effect of three different beta-glucans in combination with two probiotic strains on urate levels in faecal fermentation supernatants using stool samples from hyperuricaemic individuals | 24 hours
  Freshly collected faecal samples will be diluted and incubated with different beta-glucans and two probiotic strains for 24 hours, supernatants will be analysed for urate levels

SECONDARY OUTCOMES:
Effect of three different beta-glucans in combination with two probiotic strains on upstream and downstream metabolites of urate in faecal fermentation supernatants using stool samples from hyperuricaemic individuals | 24 hours
  Freshly collected faecal samples will be diluted and incubated with different beta-glucans and two probiotic strains for 24 hours, supernatants will be analysed for urate levels
Effect of three different beta-glucans in combination with two probiotic strains on on short-chain fatty acids (SCFA) in faecal fermentation supernatants using stool samples from hyperuricaemic individuals | 24 hours
  Freshly collected faecal samples will be diluted and incubated with different beta-glucans and two probiotic strains for 24h, supernatants will be analysed for short-chain fatty acids (SCFA)

OTHER OUTCOMES:
Effect of three different beta-glucans in combination with two probiotic strains on general microbial activity (e.g., pH) of the faecal fermentation extracts using stool samples from hyperuricaemic individuals | 24 hours
  Freshly collected faecal samples will be diluted and incubated with different beta-glucans and two probiotic strains for 24h, supernatants will be analysed for general microbial activity (e.g., pH)
Effect of three different beta-glucans in combination with two probiotic strains on the faecal microbiome of the faecal fermentation extracts using stool samples from hyperuricaemic individuals | 24 hours
  Freshly collected faecal samples will be diluted and incubated with different beta-glucans and a probiotic product, and the faecal microbiome will be analysed in the pellets (by sequencing)
Effect of three different beta-glucans in combination with two probiotic strains on the metagenetic activity (using transcriptomics) of the faecal fermentation extracts using stool samples from hyperuricaemic individuals | 24 hours
  Freshly collected faecal samples will be diluted and incubated with different beta-glucans and a probiotic product for 24h, pellets will be analysed regarding metagenetic activity (from transcriptomics)
Effect of three different beta-glucans in combination with two probiotic strains on the metagenetic activity (using metabolomics) of the faecal fermentation extracts using stool samples from hyperuricaemic individuals | 24 hours
  Freshly collected faecal samples will be diluted and incubated with different beta-glucans and two probiotic strains for 24h, pellets will be analysed regarding metagenetic activity (from metabolomics) using stool samples from hyperuricaemic individuals
Combined data analysis to explore potential responders/non-responder characteristics to treatment with a probiotic product with or without beta-glucans | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No